CLINICAL TRIAL: NCT04193111
Title: Validation of the Screening Questionnaire for Pain Attributed to Temporomandibular Disorders of Danish Headache Patients
Brief Title: Validation of the TMD Pain Screener in a Specialized Headache Center
Status: Completed | Type: Observational
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Henrik Schytz, Chief medical officer, associate professor, MD, PhD, Danish Headache Center
Other Study IDs: 061219
Record Dates: First submitted 2019-12-06; First posted 2019-12-10 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Temporomandibular Disorder; Headache Disorders
Keywords: orofacial pain; DC/TMD
MeSH Terms: conditions — Temporomandibular Joint Disorders; Headache Disorders; Facial Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Positive TMD pain screener: Patients who have ≥3 points on the TMD pain screener (0-7 range) are anticipated to have a painful TMD based on the DC/TMD and are therefore considered having a positive outcome on the TMD pain screener.
  Interventions: Diagnostic Test: TMD pain screener
- Negative TMD pain screener: Patients who have <3 points on the TMD pain screener (0-7 range) are anticipated NOT to have a painful TMD based on the DC/TMD and are therefore considered having a negative outcome on the TMD pain screener.
  Interventions: Diagnostic Test: TMD pain screener

INTERVENTIONS:
Diagnostic Test: TMD pain screener — The danish TMD pain screener is given to all participants

SUMMARY:
The purpose of the study is to investigate whether a questionnaire can be used to detect whether patients referred to the Danish Headache Center have a painful temporomandibular disorder (TMD).

TMD is a major public health problem that affects up to 15% of the adult population and can cause headaches that can be immediately difficult to differentiate from other headache types such as tension headaches and migraines. By applying the so-called diagnostic criteria for TMD through a standardized study program, TMD diseases such as myalgia of the jaw muscles, arthralgia and discus displacements of the jaw joints and jaw arthritis can be diagnosed. However, this requires dental expertise and is time consuming. At the Danish Headache Center, the current screening question is used for TMD in order to identify who could benefit from further investigation in dentistry. But it is still unknown how accurate these questions are in selecting those patients who have TMD diseases in a patient group with a headache. The investigators would like to investigate this in order to improve the referral procedure of headache patients for relevant dental treatment or physiotherapy. This is believed to be of importance both in a specialized unit such as the Danish Headache Center and in neurological medical practice.

Patients will be recruited who are referred to the Danish Headache Center, who have been given TMD screening questions and who have indicated in writing that they wish to be contacted for research projects.

In the study, 25 subjects with TMD screening question score of ≥ 3 points will be included, which will be gender and age matched with 25 subjects who have TMD screening question score of <3 points. The patients will be interviewed to classify the patients headache 15 min and then have a jaw examination done and then the DC / TMD examination will be done and lasts approx. 30 min. The examination is performed by a skilled physiotherapist and it does not involve any side effects or risks.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 18 and 75 who are referred to the Danish Headache Center

Exclusion Criteria:

* No known pre-existing significant TMD or dental disease that can cause headaches
* Anamnestic or clinical signs of a condition of any kind that is considered relevant by the investigating physician for participation in the study.
* Patients who do not wish to be informed of the findings of presence of TMD

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients referred to the Danish Headache Center with any type of headache are included. Half the population has a high probability of having a painful TMD, the other half is matched on age and gender but has a low probability of having a painful TMD.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2020-01-28 (Actual); Study Completion 2020-01-28 (Actual)

PRIMARY OUTCOMES:
Diagnostic Accuracy | baseline
  Agreement on diagnoses expressed with sensitivity and specificity

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Winther Schytz, MD, PhD, Principal Investigator — Danish Headache Center
Locations (1):
- Danish Headache Center Rigshospitalet - Glostrup, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available

REFERENCES:
- [Background] List T, Jensen RH. Temporomandibular disorders: Old ideas and new concepts. Cephalalgia. 2017 Jun;37(7):692-704. doi: 10.1177/0333102416686302. Epub 2017 Jan 9. PMID 28068790
- [Background] Adern B, Minston A, Nohlert E, Tegelberg A. Self-reportance of temporomandibular disorders in adult patients attending general dental practice in Sweden from 2011 to 2013. Acta Odontol Scand. 2018 Oct;76(7):530-534. doi: 10.1080/00016357.2018.1487076. Epub 2018 Jun 22. PMID 29932779
- [Background] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949
- [Background] List T, Ekberg C, Ernberg M, Svensson P, Alstergren P. Ny diagnostik för de vanligaste temporomandibulära dysfunktionerna för användning i allmäntandvården. Tandlægebladet 215; 119:268-276.
- [Background] Schiffman E, Ohrbach R, Truelove E, Look J, Anderson G, Goulet JP, List T, Svensson P, Gonzalez Y, Lobbezoo F, Michelotti A, Brooks SL, Ceusters W, Drangsholt M, Ettlin D, Gaul C, Goldberg LJ, Haythornthwaite JA, Hollender L, Jensen R, John MT, De Laat A, de Leeuw R, Maixner W, van der Meulen M, Murray GM, Nixdorf DR, Palla S, Petersson A, Pionchon P, Smith B, Visscher CM, Zakrzewska J, Dworkin SF; International RDC/TMD Consortium Network, International association for Dental Research; Orofacial Pain Special Interest Group, International Association for the Study of Pain. Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) for Clinical and Research Applications: recommendations of the International RDC/TMD Consortium Network* and Orofacial Pain Special Interest Groupdagger. J Oral Facial Pain Headache. 2014 Winter;28(1):6-27. doi: 10.11607/jop.1151. PMID 24482784